CLINICAL TRIAL: NCT02920502
Title: Effect of a One Time Dose of Cholecalciferol on Serum Concentration of 25-Hydroxyvitamin D and Macrophages
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Kurt Lu, Assistant Professor, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-13-15
Record Dates: First submitted 2016-09-09; First posted 2016-09-30 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1: Placebo (Placebo Comparator): Normal Healthy Volunteers without any skin pathology, will receive placebo
  Interventions: Other: Arm 1: Placebo
- Arm 2: cholecalciferol: 50,000 IU (Experimental): Normal healthy Volunteers will randomized into one of three groups and receive a one time dose of cholecalciferol at 50,000 IU.
  Interventions: Dietary Supplement: Arm 2: cholecalciferol 50,000 IU
- Arm 3: cholecalciferol: 100,000 IU (Experimental): Normal healthy volunteers will randomized into one of three groups and receive a one time dose of cholecalciferol at 100,000 IU.
  Interventions: Dietary Supplement: Arm 3: cholecalciferol 100,000 IU
- Arm 4: cholecalciferol: 200,000 IU (Experimental): Normal Healthy volunteers will randomized into one of three groups and receive a one time dose of cholecalciferol at 200,000 IU.
  Interventions: Dietary Supplement: Arm 4: cholecalciferol 200,000 IU

INTERVENTIONS:
Dietary Supplement: Arm 2: cholecalciferol 50,000 IU — One time dose of cholecalciferol 50,000 IU
  Arms: Arm 2: cholecalciferol: 50,000 IU
Dietary Supplement: Arm 3: cholecalciferol 100,000 IU — One time dose of cholecalciferol 100,000 IU
  Arms: Arm 3: cholecalciferol: 100,000 IU
Dietary Supplement: Arm 4: cholecalciferol 200,000 IU — One time dose of cholecalciferol 200,000 IU
  Arms: Arm 4: cholecalciferol: 200,000 IU
Other: Arm 1: Placebo — One time dose of Placebo
  Arms: Arm 1: Placebo

SUMMARY:
Optimal Vitamin D dosing to obtain adequate serum concentrations of 25-hydroxyvitamin D (25OHD) is controversial. The optimal dose and dosing interval is unknown, and the tendency over the last few years is to give higher, less frequent doses. Disease-specific dosing is of interest, and there may be optimal serum concentration targets based on disease process. The best evidence so far is for optimal bone health, where most experts agree that 25OHD serum concentration should be above 30 ng/ml.

There is mounting evidence that Vitamin D therapy will reduce inflammatory response and macrophage activation. The optimal dosing needed to decrease the inflammatory response is unclear, although our recent mouse model has demonstrated that a onetime high dose is effective. The investigators therefore hypothesize that a one-time high dose of cholecalciferol will be effective in suppression of macrophage production of tumor necrosis factor-alpha (TNFa) and inducible nitric oxide synthase (iNOS). The purpose of this pilot study is to assess the optimum dosage for the most macrophage suppression.

DETAILED DESCRIPTION:
3.4.1 Study Medication (Vitamin D/Placebo): Patients will be blocked randomized into one of four groups using a balanced assignment. The target number of patients is 20, with five patients who have successfully completed all assessments in each group. Groups will be closed to enrollment once their target is reached. The recruitment will continue until every group has reached its target. The investigative pharmacy will prepare each dosage according to the randomization and will hold the key to the dosing.

Participants and investigators will be blinded to those receiving cholecalciferol which comes in 50,000 I.U. dose capsules and those receiving a placebo. Participants will be randomized to 1 of 4 doses as outlined below. All participants will receive the same number of capsules. Five participants will be in each group and will be dosed according to the following dosing schema:

Table 1: Dosing Schema

Cholecalciferol Dosage Group

Control: 0 Cholecalciferol Capsules 4 Placebo Capsules

50,000 I.U.: 1 Cholecalciferol Capsules 3 Placebo Capsules

100,000 I.U.: 2 Cholecalciferol Capsules 2 Placebo Capsules

200,000 I.U.: 4 Cholecalciferol Capsules 0 Placebo Capsules

3.4.2. Skin Thickness Measurement:All testing sites will be evaluated for redness. Skin thickness will also be measured using a micrometer before and after UV exposure.

3.4.3. MED/Sunburn Test: This procedure involves exposing eight 6mm areas of skin over increasing doses of simulated solar radiation (SSR), while the rest of the body is draped. SSR is delivered by a 1,000-Watt xenon arc lamp, which emits ultraviolet wavelengths from 290-400 nm, closely resembling natural sunlight. The minimal erythema dose (MED) will be determined approximately 24 hours after initial exposure by using a chromameter that records the values of redness associated with each exposed 1cm area. The overall differences in MED between the subjects will be assessed.

3.4.4. UVR Exposure: This procedure involves exposing four 6mm areas of skin over increasing doses of simulated solar radiation (SSR), while the rest of the body is draped. SSR is delivered by a 1,000-Watt xenon arc lamp, which emits ultraviolet wavelengths from 290-400 nm, closely resembling natural sunlight. The sites to be exposed will be dosed as follows: 1 MED, 2 MED, 3 MED, 3 MED. Two sites will be exposed for this study, one before study medication dosing and one after study medication dosing.

3.4.5. Blood Draw: samples will be taken by venipuncture to provide samples for analysis of serum 25OHD and macrophages.

* Serum 25OHD and 1,25(OH): Up to 6ml blood will be drawn to measure 25OHD and sent to Heartland Assays, LLC.
* Banked Serum:Up to 30ml of blood serum will be collected and stored in the Dermatology research lab and will then be analyzed with the Macrophage Harvest.
* Macrophage Harvest: One-time collection up to 180ml whole blood will be processed and purified to isolate peripheral blood macrophages in the Dermatology research lab.

3.4.6. Punch Biopsy (Tissue Sample): A punch biopsy is the removal of a small (pencil eraser-sized) circle of skin using a cookie cutter-like instrument. This procedure involves numbing the designated area of skin with lidocaine and the removal of a circle of skin. Prior to obtaining the punch biopsy, the skin will be injected with lidocaine, a painkiller similar to that used by dentists. Although the lidocaine can tingle or hurt briefly during the numbing process, volunteers should not feel any pain while the punch biopsy is being obtained. The circle is then closed using one to five fine stitches per site, which prevents bleeding, speeds healing, and improves the appearance. The stitches are removed 10-14 days later.

3.4.7. Photographs: Photographs of the testing sites will be taken through-out this protocol. In the event that a photograph is taken of the subject's face or any other identifiable feature, the subject's identity may become known.

3.5. STUDY VISITS

3.5.1 Screening Visit

* Informed Consent
* Inclusion and Exclusion Criteria
* Medical & Dermatological History
* Physical Examination and Vital Signs of Concomitant Medications/Procedures
* Blood Draw: baseline serum vitamin D levels and banked serum
* Photographs of testing sites of MED testing

3.5.2 Visit 2: UVR #1

* Review of Inclusion and Exclusion Criteria
* Review of Adverse Events & Concomitant Medications/Procedures of chromameter reading
* Photographs of testing sites
* Site #1 UVR Exposure: 1, 2, 3, and 3 MED

3.5.3 Visit 3: 24hours post UVR #1

* Review of Inclusion and Exclusion Criteria
* Review of Adverse Events & Concomitant Medications/Procedures
* Chromameter reading
* Photographs of testing sites
* Skin Thickness Measurements

3.5.4 Visit 4: 48 hours post UVR #1

* Review of Inclusion and Exclusion Criteria
* Review of Adverse Events & Concomitant Medications/Procedures of chromameter reading
* Photographs of testing sites
* Skin Thickness Measurements
* Punch Biopsy of one 3 MED from site #I

3.5.5 Visit 5: 72 hours post UVR #1

* Review of lnclusion and Exclusion Criteria
* Review of Adverse Events & Concomitant Medications/Procedures of chromameter reading
* Photographs of testing sites
* Skin Thickness Measurements

3.5.6 Visit 6:1week post UVR #1

* Review of lnclusion and Exclusion Criteria
* Review of Adverse Events & Concomitant Medications/Procedures of chromameter reading
* Photographs of testing sites
* Skin Thickness Measurements

3.5.7 Visit 7: UVR #2: 2 weeks post UVR #1

* Review of lnclusion and Exclusion Criteria
* Review of Adverse Events & Concomitant Medications/Procedures of Photographs of testing sites
* Skin Thickness Measurements
* Site #2 UVR Exposure: I, 2, 3, and 3 MED
* One-time dose of study medication (vitamin D or placebo), 1 hour after UVR

3.5.8 Visit 8: 24 hours post UVR #2

* Review of lnclusion and Exclusion Criteria
* Review of Adverse Events & Concomitant Medications/Procedures of Chromameter reading
* Photographs of testing sites
* Skin Thickness Measurements
* Blood Draw: Serum vitamin D levels and banked serum

3.5.9 Visit 9: 48 hours post UVR #2

* Review of lnclusion and Exclusion Criteria
* Review of Adverse Events & Concomitant Medications/Procedures of chromameter reading
* Photographs of testing sites
* Skin Thickness Measurements
* Blood Draw: Serum vitamin D levels and banked serum
* Punch Biopsy of one 3 MED from site #2

3.5.10 Visit 10: 72 hours post UVR #2

* Review of Inclusion and Exclusion Criteria
* Review of Adverse Events & Concomitant Medications/Procedures
* Chromameter reading
* Photographs of testing sites
* Skin Thickness Measurements
* Blood Draw: Serum vitamin D levels and banked serum

3.5.11 Visit 11: 1 week post UVR #2

* Review of Inclusion and Exclusion Criteria
* Review of Adverse Events & Concomitant Medications/Procedures of chromameter reading
* Photographs of testing sites
* Skin Thickness Measurements
* Blood Draw: Serum vitamin D levels and banked serum

3.5.12 Visit 12: 2 weeks post UVR #2

* Review of Inclusion and Exclusion Criteria
* Review of Adverse Events & Concomitant Medications/Procedures of chromameter reading
* Photographs of testing sites
* Skin Thickness Measurements
* Blood Draw: Serum vitamin D levels and banked serum

3.5.13 Visit 13: One month post UVR #2

* Review of Inclusion and Exclusion Criteria
* Review of Adverse Events & Concomitant Medications/Procedures
* Photographs of testing sites

  4. RISKS AND DISCOMFORTS - MINIMIZED

4.1. Study Medication (Vitamin D/Placebo): Vitamin D is well tolerated and often used in clinical practice. It is freely available as an over the counter supplement. There are few side effects to oral vitamin D, with the most severe being hypercalcemia with prolonged use of a high dose. Vitamin D toxicity can occur when the active form is given (1,25 dihydroxyvitamin D) or with prolonged exposure to high dose vitamin D3. Both young and old adults have taken one time high dose vitamin D3 safely. It is possible that an allergic reaction could occur to the medication and participants will be asked to report and symptoms.

4.2. Skin Thickness Measurement: there are no known risks to evaluating or measuring the skin's thickness with a micrometer.

4.3. Minimal Erythema Dose (MED) and Ultraviolet Light Exposure (UVR): The risks associated with this procedure are minimal, as only the testing sites will be exposed. The consequences of being exposed to UV light are short-term, and primarily involve mild redness at the exposure site followed by minor itching and dryness of the skin several days later. The degree of the sunburn is typically mild to moderate and the UV dose used is not enough to cause blistering of the skin.

4.4. Blood Draw: Risks from a blood draw may include the occurrence of discomfort and/or bruise at the site of puncture and, less likely, the formation of a small clot, swelling of the vein, or bleeding from the puncture site.

4.5. Punch Biopsy (Tissue Sample): Punch biopsies pose minimal risk, and volunteers are instructed as to the proper care of the biopsy site. Lidocaine may cause a tingling or burning sensation when injected into the skin. Potential problems localized to the biopsy site include bleeding or oozing, discomfort, or infection. The biopsy site will heal with a small, flat scar, which may be red for several months. The scar may also turn lighter or darker than the surrounding skin after some time.

4.6. Photographs: There are no known risks to taking photographs. In the event a photograph is taken of the subject's face or any other identifying feature, the patient's identity may be known.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18 years or older
* Fitzpatrick Skin Type I-Ill
* In good general health and able to list all current medications and medical conditions
* Capable of giving informed consent

Exclusion Criteria:

* Volunteers ages 18 years or younger
* Women who are pregnant, nursing, or who may become pregnant in the next 3 months
* Participants taking illegal drugs
* Chronic medical conditions
* Currently taking statins, ketoconazole, colestipol, cholestyramine, phenobarbitol, phenytoin, or mineral oil
* Currently consuming 800 IU or more of vitamin D a day
* Current or recent use of anti-inflammatory medications or any other medications that may cause photosensitivity, at the discretion of the Pl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Primary Measure Assessing Change of Erythema and Edema | 24 hours, 48 hours, 72 hours, 1 week, 2 weeks
  MED testing & Recovery from UV-induced erythema and edema before a one time dose of cholecalciferol

SECONDARY OUTCOMES:
Secondary Measure Assessing Change of Serum Vitamin D Levels and Skin Inflammation | Before:24 hours, 48 hours, 72 hours, 1 week, 2 weeks ; After: 24 hours, 48 hours, 72 hours, 1 week, 2 weeks, 1 month
  Sample Analysis (from blood and skin): Skin and blood samples will be collected from all study subjects to look at serum vitamin D levels and the effect of serum 25OHD concentration on levels of pro-inflammatory factors in the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Lu, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heaney RP, Armas LA, Shary JR, Bell NH, Binkley N, Hollis BW. 25-Hydroxylation of vitamin D3: relation to circulating vitamin D3 under various input conditions. Am J Clin Nutr. 2008 Jun;87(6):1738-42. doi: 10.1093/ajcn/87.6.1738. PMID 18541563
- [Background] Sanders KM, Stuart AL, Williamson EJ, Simpson JA, Kotowicz MA, Young D, Nicholson GC. Annual high-dose oral vitamin D and falls and fractures in older women: a randomized controlled trial. JAMA. 2010 May 12;303(18):1815-22. doi: 10.1001/jama.2010.594. PMID 20460620
- [Background] van Groningen L, Opdenoordt S, van Sorge A, Telting D, Giesen A, de Boer H. Cholecalciferol loading dose guideline for vitamin D-deficient adults. Eur J Endocrinol. 2010 Apr;162(4):805-11. doi: 10.1530/EJE-09-0932. Epub 2010 Feb 5. PMID 20139241